CLINICAL TRIAL: NCT02908386
Title: In Silico Clinical Trial on Adaptive Radiotherapy in Oropharynx Cancer, Comparing Photon & Proton Therapy: A Multicentric ROCOCO Planning Study Based on a Reference Dataset.
Brief Title: ROCOCO - Adaptive IMRT Versus IMPT in Head and Neck Cancer
Acronym: ROCOCO
Status: Withdrawn | Type: Observational
Why Stopped: At the moment no participants are enrolled untill a new agreement is made
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 2016 ROCOCO HN
Record Dates: First submitted 2016-04-13; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and neck tumors; Proton; Photon; replanning timing
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Given the lack of evidence for the benefit of particle therapy in relevant cases, he investigators proposed an in silico trial to investigate the dosimetric effect of contour changes for OAR as well as tumor during chemoradiation in H&N patients. Photon and proton-therapy will be compared based on dosimetric data on 7 time points during treatment combined with plan robustness. In that way the investigators will be able to assess and compare the optimal timing for replanning for photon and proton therapy.

A database of the University of Pennsylvania (Upenn) consists of 10 patients with head and neck tumors treated with chemo-radiation. Contrast-enhanced CT scans were acquired prior and during RT (T1-T7)

DETAILED DESCRIPTION:
Given that the cost of particle therapy (PT) is considerably higher than that of conventional radiotherapy (RT) with photons, it is necessary to establish whether these higher costs are worthwhile in light of the expected advantages. Thus, clear evidence of the situations in which PT outperforms conventional photon treatment is needed. ROCOCO (Radiation Oncology COllaborative Comparison) is commenced at MAASTRO in May 2007 to evaluate PT's cost-effectiveness .

It is well known that during radiation treatment of head and neck cancer (HN), shrinkage and displacement of tumour and organs at risk (OARs, e.g. parotid glands), as well as weight loss may cause significant radiation dose changes to target volumes and organs at risk , , . These phenomena may cause the necessity to re-plan the treatment at a certain moment in time. In the last years many different treatment planning studies have been performed showing that the optimum moment for re-planning varies: after 20 Gy, 35 or 46 Gy. But what the actual effect of the deformation is on dose in actually treated patients has not been reported.

The investigators propose an in silico trial to investigate the relevance of contour changes for OAR as well as tumor during chemo radiation in H&N patients which will eventually lead to replanning. In that way the investigators will be able to assess and compare the optimal timing for replanning for photon and proton therapy.

The investigators compare different treatments focusing on the effect of deformation on PTV coverage and normal tissue radiation exposure. A fixed tumor dose, using the same delineation of gross target volume (GTV), clinical target volume (CTV) is used. The planning target volume (PTV) will be determined by each treatment modality.

For the initial plan the best possible dose distribution will be determined using the planning-CT (reference scan). For every time point (CT-scan) the reference treatment plan will be projected on the actual CT scan and the dose will be recalculated without changing the treatment parameters. This will be done using both photons and protons. All treatment uncertainties including robustness will be taken into account. Dose differences in the target volume (CTV-GTV and PTV) and the OAR, as a result of tumor shrinkage during treatment will be evaluated for each time point and each treatment modality.

The objective of this study is to assess plan robustness and the optimal timing for replanning for photon and proton therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with head and neck carcinoma who have been treated with radical intent 10 patients, all with a reference CT scan and CT scans at 7 time points during treatment.

Exclusion Criteria:

* patients with no head and neck cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 10 consecutive patients treated with proton therapy at the University of Pennsylvania (USA). Other treatment modalities for the tumor sites, such as chemotherapy will not be taken into account. Included are H&N patients who have been treated with radical intent. Each patient will function as his or her own control.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Dose distribution | up to 26 weeks
  Dose values of seven time frames (T1-T7) are compared to the reference dose values on the planning CT for both photon and proton treatment plans.

SECONDARY OUTCOMES:
Optimal timing for replanning | up to 26 weeks
  Determine the optimal timing for replanning for each modality when taking all the treatment uncertainties in account.

OTHER OUTCOMES:
Plan uncertainties and robustness | up to 26 weeks
  Investigate plan uncertainties and robustness for photon and proton therapy in adaptive H&N tumors

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, Prof dr, Study Director — Maastro Clinic, The Netherlands
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Roelofs E, Engelsman M, Rasch C, Persoon L, Qamhiyeh S, de Ruysscher D, Verhaegen F, Pijls-Johannesma M, Lambin P; ROCOCO Consortium. Results of a multicentric in silico clinical trial (ROCOCO): comparing radiotherapy with photons and protons for non-small cell lung cancer. J Thorac Oncol. 2012 Jan;7(1):165-76. doi: 10.1097/JTO.0b013e31823529fc. PMID 22071782
- [Result] Barker JL Jr, Garden AS, Ang KK, O'Daniel JC, Wang H, Court LE, Morrison WH, Rosenthal DI, Chao KS, Tucker SL, Mohan R, Dong L. Quantification of volumetric and geometric changes occurring during fractionated radiotherapy for head-and-neck cancer using an integrated CT/linear accelerator system. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):960-70. doi: 10.1016/j.ijrobp.2003.12.024. PMID 15234029
- [Result] Ricchetti F, Wu B, McNutt T, Wong J, Forastiere A, Marur S, Starmer H, Sanguineti G. Volumetric change of selected organs at risk during IMRT for oropharyngeal cancer. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):161-8. doi: 10.1016/j.ijrobp.2010.01.071. Epub 2010 Nov 19. PMID 21306971
- [Result] Geets X, Tomsej M, Lee JA, Duprez T, Coche E, Cosnard G, Lonneux M, Gregoire V. Adaptive biological image-guided IMRT with anatomic and functional imaging in pharyngo-laryngeal tumors: impact on target volume delineation and dose distribution using helical tomotherapy. Radiother Oncol. 2007 Oct;85(1):105-15. doi: 10.1016/j.radonc.2007.05.010. Epub 2007 Jun 11. PMID 17562346